CLINICAL TRIAL: NCT02647905
Title: A Prospective, Multicenter Evaluation of the Accuracy of a Novel Continuous Implanted Glucose Sensor, PRECISE II
Brief Title: Evaluation of the Accuracy of an Implanted Glucose Sensor
Acronym: PRECISEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0023
Record Dates: First submitted 2015-12-31; First posted 2016-01-06 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus
Keywords: type 1 diabetes; type 2 diabetes; CGM; implantable; accuracy; longevity
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accuracy assessment, CGMS (Experimental): To determine accuracy of the Senseonics Continuous Glucose Monitoring System measurements through approximately 90 days post-insertion. Manipulation of glucose levels during multiple clinic days
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Accuracy and safety assessment of a continuous glucose monitoring device

SUMMARY:
The purpose of this clinical investigation is to evaluate the accuracy of the Senseonics Continuous Glucose Monitoring System (Senseonics CGM System) measurements when compared with reference standard measurements The investigation will also evaluate safety of the Senseonics CGM System usage.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, age ≥18 years
2. Clinically confirmed diagnosis of diabetes mellitus for ≥1 year
3. Subject has signed an informed consent form and is willing to comply with protocol requirements

Exclusion Criteria:

1. History of severe hypoglycemia in the previous 6 months. Severe hypoglycemia is defined as hypoglycemia resulting in loss of consciousness or seizure
2. History of diabetic ketoacidosis requiring emergency room visit or hospitalization in the previous 6 months
3. Female subjects of childbearing capacity (defined as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study.
4. A condition preventing or complicating the placement, operation, or removal of the Sensor or wearing of transmitter, including upper extremity deformities or skin condition.
5. Symptomatic coronary artery disease; unstable angina; myocardial infarction, transient ischemic attack or stroke in the past 6 months; uncontrolled hypertension (systolic>160 mm Hg or diastolic >100 mm Hg at time of screening); current congestive heart failure; history of cardiac arrhythmia (benign PACs and PVCs allowed). Subjects with asymptomatic coronary artery disease (e,g, CABG, stent placement or angioplasty) may participate if negative stress test within 1 year prior to screening and written clearance from Cardiologist documented.
6. Hematocrit <30% or >55%
7. History of hepatitis B, hepatitis C, or HIV
8. Any condition that in the investigator's opinion would make the subject unable to complete the study or would make it not in the subject's best interest to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research
Locations (9):
- United States (9):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Care, Atlanta, Georgia
  - Mount Sinai Diabetes Center, New York, New York
  - Worldwide Clinical Trials, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - UVA Diabetes and Endocrine Clinic, Charlottesville, Virginia
  - Rainier Clinical Research, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Accuracy Assessment, CGMS
Started | 90
Completed | 87
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Accuracy Assessment, CGMS
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 77
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90
Dominant Hand [Count of Participants; unit: Participants]
  Right | 78
  Left | 12
Body mass Index [Count of Participants; unit: Participants]
  Normal (<25 kg/m2) | 22
  Overweight (≥25 and <30) | 27
  Obese (≥ 30) | 41
Years since diabetes diagnosis [Mean (Standard Deviation); unit: years] | 20.1 (13.7)
Diabetes Type [Count of Participants; unit: Participants]
  Type I | 61
  Type II | 29
Type of insulin therapy [Count of Participants; unit: Participants]
  None | 20
  Multiple daily injections | 24
  continuous insulin infusion pump | 43
  Other | 3
History of [Count of Participants; unit: Participants]
  Ketoacidosis | 0
  Hypoglycemia | 1

OUTCOME MEASURES:

1. Primary Outcome: CGM Relative Difference to Laboratory Reference Reported as MARD
Description: Mean absolute relative difference (MARD) for paired Sensor and reference measurements through 90 days post-insertion for reference glucose values from 40-400 mg/dL will be calculated for comparison.
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Accuracy Assessment, CGMS
Number analyzed (Participants) | 87
percent | 8.5 [8.0 to 9.1]

2. Other Pre Specified Outcome: CGM System Agreement With Reference Control
Description: The percentage of system readings within ±15 mg/dL or 15% of YSI reference values (15/15%)
Time Frame: 90 days
Measure: Number; unit: percent of readings within 15/15%
Arm/Group | Accuracy Assessment, CGMS
Number analyzed (Participants) | 87
percent of readings within 15/15% | 86.8

ADVERSE EVENTS:
Time Frame: 90 days post insertion or sensor removal and follow-up
Arm/Group | Accuracy Assessment, CGMS
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 1/90
Other Adverse Events (participants affected / at risk) | 43/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accuracy Assessment, CGMS (N=90)
Surgical procedure to remove sensor (Surgical and medical procedures) | 1 (1) — PI requested assistance from a general surgeon for removal of sensor through outpatient surgery who then elected to place the patient under general anesthesia. The sensor was removed intact without incident
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accuracy Assessment, CGMS (N=90)
Food poisoning (Injury, poisoning and procedural complications) | 1 (1) — Not related to Study device or insertion/removal procedure
Syncope (Vascular disorders) | 2 (2) — Related or Possibly related to Study Procedure
Carpal tunnel (Nervous system disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Dizziness (Nervous system disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Headache (Nervous system disorders) | 4 (5) — Related or Possibly related to Study Procedure
Paresthesia (Nervous system disorders) | 1 (1) — Related or Possibly related to the study device or Insertion/Removal Procedure
Syncope-Vasovagal (Vascular disorders) | 1 (1) — Related or Possibly related to the study device or Insertion/Removal Procedure
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Not related to Study device or insertion/removal procedure
Neck strain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Broken toe (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Rib injury (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Sensor location site- Pain/discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) — Related or Possibly related to the study device or Insertion/Removal Procedure
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Nephrolithiasis (Renal and urinary disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Candidiasis vaginal (Reproductive system and breast disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Dyslipidemia (Metabolism and nutrition disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Fever (General disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Common cold (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Not related to Study device or insertion/removal procedure
Sore throat (Gastrointestinal disorders) | 2 (2) — Not related to Study device or insertion/removal procedure
Cracked tooth (Injury, poisoning and procedural complications) | 1 (1) — Not related to Study device or insertion/removal procedure
Infection-Tooth (Infections and infestations) | 1 (1) — Not related to Study device or insertion/removal procedure
Laryngitis (Infections and infestations) | 1 (1) — Not related to Study device or insertion/removal procedure
Cataracts (Eye disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Infection-Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Blepharoplasty (Surgical and medical procedures) | 1 (1) — Not related to Study device or insertion/removal procedure
Broken tooth (Injury, poisoning and procedural complications) | 1 (1) — Not related to Study device or insertion/removal procedure
TMJ pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Device Fragement not recovered (Surgical and medical procedures) | 2 (2) — Related or Possibly related to the study device or Insertion/Removal Procedure
Fatigue (General disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Bruising (Skin and subcutaneous tissue disorders) | 1 (2) — Related or Possibly related to the study device or Insertion/Removal Procedure
Erythema, removal site (Skin and subcutaneous tissue disorders) | 1 (2) — Related or Possibly related to the study device or Insertion/Removal Procedure
Sensor location site- Pain/discomfort (General disorders) | 3 (4) — Related or Possibly related to the study device or Insertion/Removal Procedure
IV site pain (Injury, poisoning and procedural complications) | 1 (1) — Related or Possibly related to Study Procedure
Dermatitis (Immune system disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Cellulitis (Infections and infestations) | 1 (1) — Not related to Study device or insertion/removal procedure
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
IV site Erythema (Injury, poisoning and procedural complications) | 1 (1) — Related or Possibly related to Study Procedure
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Gastroenteritis (Gastrointestinal disorders) | 4 (4) — Not related to Study device or insertion/removal procedure
Constipation (Gastrointestinal disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Gastric ulcer (Gastrointestinal disorders) | 1 (1) — Not related to Study device or insertion/removal procedure
Diarrhea (Gastrointestinal disorders) | 2 (2) — Not related to Study device or insertion/removal procedure
Nausea (Gastrointestinal disorders) | 2 (2) — Not related to Study device or insertion/removal procedure
Erythema, Arm (Skin and subcutaneous tissue disorders) | 1 (1) — Related or Possibly related to Study Procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less